CLINICAL TRIAL: NCT00521768
Title: Effectiveness of Prolonged Exposure of PTSD in a Community Setting of PTSD Sufferers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT20
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Post Traumatic Stress Disorder; Anxiety Disorder
Keywords: Post traumatic stress disorder; Anxiety disorder; Comunity base intervention; Education; Behavioural treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders

INTERVENTIONS:
Behavioral: Prolonged exposure

SUMMARY:
Introduction: Efforts to bridge the gap between research based treatment modalities advancements and clinical practice have received the highest priority in the research community. In the child psychiatry field there is an urging need to promote bridging this gap.

Parents and child health providers hesitate to refer children to child psychiatrist due to stigma but also due to lack of awareness of available and efficient treatment options. In the field of trauma treatment another reason for lack of treatment is lack of recognition of trauma related symptoms in children.

After the second Lebanon war scarce referrals to psychiatric clinics have been registered and access to treatment is low as indicated by 20 referrals in the past year to Emek Hospital.

We propose to explore the effectiveness of well-established adult treatment for PTSD, the Prolonged Exposure (PE), in community-based general pediatric clinics, serving an underprivileged diverse population.

Methods:

Twenty children age 6 to 18 attending general pediatric clinic and in Afula region will included.

children will be diagnosed using the Hebrew translation of the Childhood version of the Schedule for Affective Disorders and Schizophrenia (Apter et al., 1989 Children will receive the Children's Depression Inventory (CDI) and the. CPSS All subjects will be treated with a manualized 12-week Prolonged Exposure protocol Ratings will be made at baseline, 6weeks, and 12 weeks using CDI and CPSS

Hypothesis:

1. PE adapted for pediatric population will be effective in treating single-event traumas in a community setting.

DETAILED DESCRIPTION:
SPECIFIC AIMS The aim of the study is to examine the effectiveness of PE treatment of PTSD in community settings

BACKGROUND AND SIGNIFICANCE There is a great need to apply scientific achievements in behavioral science research to community-based clinical settings. Many recent advances in psychology with significant potential to improve clinical practice and intervention have not yet been utilized in clinical settings.

A recent report of the NIH National Advisory Mental Health Council Behavioral Science Workgroup has defined this approach, "Translational research", as follows: "Translational research in the behavioral and social sciences addresses how basic behavioral processes inform the diagnosis, prevention, treatment and delivery of services for mental illness, and conversely, how knowledge of mental illness increases our understanding of basic behavioral processes. " (NIH publication, 2001).

PTSD in children is a well established diagnosis.Recent studies have shown 30 % of children presenting with PTSD symptoms after the second Lebanon war Parents and child health providers hesitate to refer children to child psychiatrist due to stigma but also due to lack of awareness of available and efficient treatment options. In the field of trauma treatment another reason for lack of treatment is lack of recognition of trauma related symptoms in children.

After the second Lebanon war scarce referrals to psychiatric clinics have been registered and access to treatment is low as indicated by 20 referrals in the past year to Ha'Emek Medical Center child and adolescent psychiatric clinic.

Ha'Emek medical center is initiating a community base PTSD treatment program to children attending general pediatric clinics.

We propose to explore the effectiveness of well-established adult treatment for PTSD, the Prolonged Exposure (PE), in community-based general pediatric clinics, serving an underprivileged diverse population.

RESEARCH DESIGN AND METHODS Subjects: Twenty children age 6 to 18 referred to the community base PTSD treatment program offered by the Ha'Emek medical center in Afula will be include: All families referred to the PTSD treatment program will be offered to participate in the research protocol. We expect 50 families to be included in the treatment program. Only subject whose both parents will agree for inclusion in the research program will be included.

DSM- IV R diagnosis: PTSD Evaluation/Instruments Socio-Demographics Data: Child: Age, Sex, grade level and medical history. Parents: Age, marital status, ethnic background, country of birth, language spoken at home, education level, occupational status.

Trauma History: Type of trauma, distance from Katushe fall Kiddy SADS: a semi structural interview CDI: a self report questionnaire CPSS: a self report questionnaire

Procedures:

Parents will be informed of the goals of the study by their primary child health provider, and will be offered the opportunity to meet with the mental health worker prior to enrollment.. Parents will be told that their participation in the research is voluntary and anonymous and their refusal to participate will not affect the services they receive by the project.

Children who will be diagnosed as having PTSD will be offered 12 sessions treatment by PE.

CDI and CPSS will be scored at time 0, time 6 weeks and time 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Children age 6 to 18
* Language spoken: Hebrew
* DSM- IV R diagnosis: PTSD
* Anxiety disorder

Exclusion Criteria:

* Children presenting with psychotic symptoms,
* Children presenting with mental retardation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
CDI questionaire | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Bracha, MD, Principal Investigator — HaEmek MC
Locations (1):
- HaEmek Medical Center - Psychiatry Department, Afula, Afula, Israel